CLINICAL TRIAL: NCT03675490
Title: ABLE (Arts-Based Exercise Enhancing LongEvity): Interactive, Arts-based Technology to Support Sustainable Exercise Participation in the Homes of Older Adults: Protocol for a Pre-post Pilot Feasibility Study
Brief Title: ABLE (Arts-Based Exercise Enhancing LongEvity)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: McMaster Institute for Research on Aging (Unknown); Physiotherapy Foundation of Canada (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABLEPILOT
Record Dates: First submitted 2018-09-13; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Aging; Fall; Muscle Weakness; Mobility Limitation
MeSH Terms: conditions — Muscle Weakness; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: pre-post pilot feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Participants will engage in a physiotherapist-prescribed home exercise program with ABLE, the interactive technology. The exercises that will be prescribed are designed to improve functional mobility via challenging lower extremity strength and balance in a multicomponent exercise program. The difficulty of each exercise will be chosen at the discretion of the physiotherapist based on the participants' performance on the baseline assessments. The exercises will be prescribed at a moderate intensity (moderate balance challenge, 8-12 repetitions for strength exercises with the last few repetitions being challenging) and will be progressed over the study duration to ensure they remain a moderate challenge.
  Interventions: Behavioral: ABLE - exercise with interactive technology

INTERVENTIONS:
Behavioral: ABLE - exercise with interactive technology — Multicomponent exercise with interactive technology - consists of wearable sensors and a screen displaying interaction. When the person does the exercises it produces an arts-based response on the screen (e.g., digital painting).,

SUMMARY:
Older adults who are referred to home care physiotherapy often only get to see the physiotherapist three to five times and are expected to continue exercising on their own. We have developed an interactive technology called ABLE that helps older adults do exercise in their homes by making it fun and interactive. We want to see if we can help 25 older adults to exercise with ABLE for three months and if exercising with ABLE for three months changes older adults' strength and balance. A physiotherapist will visit the older adults three times in their homes and show them how to use ABLE and which exercises to do. We will measure older adults' strength and balance before and after using the program and ask them and their family members for feedback about using ABLE. The results of our study will help us decide if we can do a bigger study to test the effect of using ABLE in a larger group of older adults, and to see what effect ABLE might have on strength and balance. The study will also help us incorporate feedback from the older adults and their families to improve ABLE for the next study.

ELIGIBILITY:
Inclusion Criteria:

* able to stand and walk independently with or without an assistive aid (e.g., walker, cane)
* may have a diagnosis of dementia or cognitive impairment (MoCA < 25, MMSE <24, Mini-Cog <3) if they have caregiver willing to assist with exercises and consent

Exclusion Criteria:

* have a diagnosis of dementia or cognitive impairment (MoCA < 25, MMSE <24, Mini-Cog <3) and have no family member to assist with exercises and consent
* documented absolute contraindications to exercise

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | One year
  The number of participants recruited over one year.
Retention | Three months
  The number of participants who complete visit 4.
Adherence | Three months
  The number of days per week that participants complete the home exercise program.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Three months
  The SPPB is a measure of lower extremity function through measures of balance (timed static stance in feet together, semi-tandem and tandem with eyes open), gait speed, and the time to rise from a chair
Balance Outcome Measure for Elder Rehabilitation (BOOMER) | Three months
  The BOOMER is a measure of static and dynamic balance
International Physical Activity Questionnaire (IPAQ) | Three months
  The IPAQ is a self-report measure of time spent (e.g., duration per session, and number of session in the past 7 days) in strength training, yoga/Tai Chi/other balance activities, vigorous physical activity, moderate physical activity, walking, and sitting/lying down while awake
Self-reported falls as reported in daily diary | Three months
  A slip or a trip where the person loses their balance and part or all of their body lands on the ground, floor, or lower level
Participant feedback | Three months
  Participants and their caregivers (if they assisted with the intervention) will provide their feedback on the technology and participation in the pilot study via one-on-one qualitative interviews completed during the last study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, MD, MSc, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: Undecided
Data available upon request.